CLINICAL TRIAL: NCT02615236
Title: Prospective Evaluation of Perineal Ultrasound in Thr Delivery Room to Improve the Diagnosis of OASIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Dr. Ahmed Kotb, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PUS-OASIS
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Episiotomy
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PERINEAL ULTRASOUND (Experimental): Perineal ultrasound with a bedside scanner by inserting a the probe into the perineum and reviewed in real-time
  Interventions: Device: perineal ultrasound
- Clinical diagnosis (Active Comparator): Diagnosis of OASIS will be clinically
  Interventions: Procedure: Clinical diagnosis

INTERVENTIONS:
Device: perineal ultrasound — transvaginal probe will be used to scan the perineum immediately after vaginal delivery in primiparous women
  Arms: PERINEAL ULTRASOUND
Procedure: Clinical diagnosis — diagnosis of OASIS clinically
  Arms: Clinical diagnosis

SUMMARY:
The aim of the study is to evaluate the role of routine perineal scan using 2D ultrasound immediatly after delivery to diagnose hidden perineal trauma that might affect patient's fecal continance

DETAILED DESCRIPTION:
In countries where there is high prevalence of doing episiotomy in primiparous women, the incidence of sustained obstetric anal sphincter injuries is increasing.

When the tear extend beyond the external anal sphincter its called 'OASIS' that might lead to either immediate of delayed anal incontinence. Anal incontinence is associated with significant medical, hygiene and social problems. Use of perineal ultrasound as a bedside test immediately after vaginal delivery could improve the diagnosis and determining the degree of these perineal traumas. This increased detection could lead to improved primary repair of the external and internal anal sphincter resulting in reduced rates of anal incontinence and improved quality of life for women

ELIGIBILITY:
Inclusion Criteria:

* primiparous women immediately after vaginal delivery

Exclusion Criteria:

* history of anal incontinence
* previous anal sphincteric injuries
* previous anal surgery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
anal incontinence | 3 months after delivery
  patients will be reviewed for anal incontinence 3 months after delivery

SECONDARY OUTCOMES:
pain score | 3 and 12 month after delivery
  visual analogue scale will be used
questionnaire for effect on quality of life | 3 and 12 month after delivery
  questionnaire will be used to asses how anal incontinence affect the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No